CLINICAL TRIAL: NCT07059988
Title: The Effect of Nutrition on Endogenous Energy Substrate Production in the Early and Late Acute Phase of Critical Illness
Brief Title: Endogenous Energy Production in Critically Ill Patients
Acronym: eEPIC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Martin Sundstrom Rehal, Principal Investigator, Karolinska University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024-9306
Record Dates: First submitted 2025-06-23; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Critical Illness; Metabolism and Nutrition Disorder
MeSH Terms: conditions — Critical Illness; Nutrition Disorders | interventions — Parenteral Nutrition

STUDY DESIGN:
Intervention Model Description: Patients and age-matched controls.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICU Patients (Experimental): Mechanically ventilated patients admitted to the study site ICU.
  Interventions: Other: Stable isotope tracers; Dietary Supplement: Parenteral nutrition
- Control group (Experimental): Non-hospitalized study subjects recruited through public advertising at the study site, age-matched on group level.
  Interventions: Other: Stable isotope tracers; Dietary Supplement: Parenteral nutrition

INTERVENTIONS:
Other: Stable isotope tracers — Deuterium-labelled non-radioactive stable isotopes of glucose, phenylalanine and glycerol.
Dietary Supplement: Parenteral nutrition — Parenteral nutrition infused a rate corresponding to 100% of measured energy expenditure, started after blood sampling during a baseline fasting period.

SUMMARY:
The aim of this study is to investigate when critically ill patients transition from a non-suppressible catabolism to a normal response to feeding.

Endogenous production of glucose, fat and protein will be studied on a minimum of two occasions in mechanically ventilated ICU patients, in a fasted state and during parenteral nutrition. Substrate kinetics are estimated by a tracer dilution method using infusions of isotopically labeled glucose, glycerol and phenylalanine. Blood sampling for metabolomics analysis will be performed to elucidate potential biomarkers indicating an anabolic response to nutrition.

DETAILED DESCRIPTION:
Background and aims

Critical illness is characterized by several metabolic alterations, including an upregulation of catabolic pathways promoting endogenous energy substrate production. In contrast to starvation catabolism, this endogenous energy supply cannot be suppressed by feeding in the early acute phase of critical illness. This observation is one of the reasons that current guidelines recommend hypocaloric nutrition during the first week in ICU [1]. However, it is not known when this anabolic resistance subsides and a transition towards a normal response to feeding occurs.

The aims of this study are two-fold: 1) to investigate the temporal changes in non-suppressible endogenous energy production during critical illness, and 2) identify potential biomarkers indicating a normalized response to exogenous nutrients.

Protocol

For ICU patients, the protocol is first performed within 24-72 hours (early acute phase) from ICU admission. The protocol will be repeated if an enrolled patient is still in the ICU 120-168 hours (late acute phase) and 240-288 hours (late phase) after the first study session.

Infusions of intravenous (i.v.) glucose, enteral/parenteral nutrition (EN/PN) and insulin are stopped at 02:00 hours. Blood glucose concentrations will be monitored at least hourly during the fasting period. The protocol will be terminated in case of hypoglycaemia (<4 mmol/L), and the patient will be excluded from the trial. The infusion rate of propofol will remain unchanged from 04:00 unless a change is clinically indicated, determined by the nurse or physician. Healthy controls will be asked to fast from midnight. In the control group, a peripheral i.v. line and a radial arterial line will be placed under local anaesthesia.

Baseline blood samples will be drawn from the arterial catheter, whereafter primed i.v. infusions of ring-2H5-phenylalanine, 2H2-glucose, and 2H5-glycerol will be started at 07:00. Measured resting energy expenditure (mREE) is then determined by 20-minute indirect calorimetry (IC) using the Q-NRG device (Cosmed, Rome, Italy) in ventilator or canopy mode. After 165 minutes, four blood samples will be drawn at 5-minute intervals from the arterial catheter to determine glucose, glycerol, and amino acid kinetics in a fasted state. Additional blood samples are drawn to analyze circulating hormones, cytokines, metabolites, and markers of autophagy.

PN (Olimel perifer N4E, Baxter) is then started at a rate that, including calories from propofol and other non-nutritional energy sources, corresponds to 100% of mREE. Repeated blood samples (same as above) are drawn at 45-60, 105-120 and 165-180 minutes after the start of PN. An additional IC is performed during the final 30 minutes of the PN. If hyperglycemia occurs during the PN administration, an insulin infusion will be started to keep blood glucose levels <14 mmol/L.

After the final blood samples, all tracer infusions and PN are stopped. In ICU patients, nutritional therapy will be restarted as prescribed by the care team. In healthy controls, all catheters are removed.

Patients

Adult patients with an estimated ICU length of stay (LOS) >72 hours will be recruited from the intensive care unit (ICU) at Karolinska University Hospital Huddinge, a tertiary university hospital with approximately 800 annual ICU admissions. Exclusion criteria include liver disease (liver transplant, acute or acute-on-chronic liver failure, cirrhosis), diabetes, pancreatic surgery or pancreatitis, pregnancy, intubation for airway protection only, mitochondrial disease, amino acid metabolism disorder, familial hypertriglyceridemia, severe hypertriglyceridaemia (≥ 10 mmol/L), hypoglycemia within the last 72 h, requiring ongoing large-volume resuscitation and/or blood transfusions, readmission within one week of ICU discharge, BMI ≥35, limitations to best supportive care or ongoing insulin/glucose treatment related to hyperkalemia.

Control group

Healthy, age- and sex-matched controls.

Statistical analysis and sample size considerations

Normal distribution will be assumed a priori. Primary and secondary outcomes will be analyzed using Student's T-test for paired or independent samples or one-way ANOVA as appropriate. The level of statistical significance is p ≤ 0.05. Correction for multiple comparisons will not be applied.

Based on previous data describing endogenous glucose production in a fasted and fed state in critically ill patients, 10 subjects in each group are required to detect a 20% difference in change in glucose rate of appearance with 80% power. No similar studies describing glycerol or amino acid kinetics are available for sample size calculations. Due to missing data, dropouts and inter-/intraparticipant variability, 10 patients with measurements of substrate kinetics in both the early acute and late acute phases are required to answer the primary and secondary outcome measures. To identify potential biomarkers of attenuated catabolism, 30 patients who complete the protocol in both the early acute and late acute phases will be included, i.e. two measurements per patient. Ten volunteers will be recruited to an age-matched control group.

ELIGIBILITY:
Inclusion Criteria:

For the ICU group:

1. ≥18 years old and admitted to the ICU
2. Invasive mechanical ventilation
3. Arterial and central line in situ
4. Expected to remain in ICU >72 hours

For the control group:

1. ≥18 years old

Exclusion Criteria:

1. Lack of informed consent by patient/next of kin
2. Liver transplant
3. Acute or acute on chronic liver failure
4. Cirrhosis
5. Known diabetes mellitus
6. Pancreatic surgery
7. Acute or chronic pancreatitis
8. Pregnancy
9. Intubated only for airway protection or neurologic deficit
10. Mitochondrial disease
11. Disorder of amino acid metabolism
12. Familial hypertriglyceridemia
13. Severe acquired hypertriglyceridemia (≥10 mmol/L)
14. Requiring treatment of hypoglycemia in the last 72 hours before inclusion.
15. Requiring ongoing large volume resuscitation of crystalloids or blood products
16. >72 hours in ICU before enrollment
17. Readmission to ICU within 1 week of ICU discharge.
18. Morbidly obese (BMI ≥35)
19. Limitations of treatment to best supportive care
20. Ongoing treatment with insulin/glucose related to hyperkalemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Attenuation of glucose production in response to nutrition in early acute phase in ICU. | Early acute phase of critical illness, i.e., 24-72 hours after ICU admission. The difference between substrate kinetics at 165-180 min and 345-360 min after the start of the tracer infusion will be calculated.
  Difference in endogenous rate of appearance of glucose, calculated from enrichment of labelled substrates in plasma of glucose between the fasted and fed state in the early acute phase in ICU.
Attenuation of phenylalanine production in response to nutrition in early acute phase in ICU. | Early acute phase of critical illness, i.e., 24-72 hours after ICU admission. The difference between substrate kinetics at 165-180 min and 345-360 min after the start of the tracer infusion will be calculated.
  Difference in endogenous rate of appearance of phenylalanine, calculated from enrichment of labelled substrates in plasma of phenylalanine, between the fasted and fed states in the early acute phase in ICU.
Attenuation of glycerol production in response to nutrition in early acute phase in ICU. | Early acute phase of critical illness, i.e., 24-72 hours after ICU admission. The difference between substrate kinetics at 165-180 min and 345-360 min after the start of the tracer infusion will be calculated.
  Difference in endogenous rate of appearance of glycerol, calculated from enrichment of labelled substrates in plasma of glycerol, between the fasted and fed states in the early acute phase in ICU.

SECONDARY OUTCOMES:
Attenuation of glucose production in response to nutrition in the late acute phase compared to the early acute phase in the ICU. | The early acute phase is between 24 and 72 hours after ICU admission, and the late acute phase between 120 and 148 hours, i.e., 5-7 days after ICU admission.
  Difference in endogenous rate of appearance, calculated from enrichment of labelled substrates in plasma glucose, between the fasted and fed state in the early acute phase, compared to the late acute phase in the ICU.
Attenuation of glycerol production in response to nutrition in the late acute phase compared to the early acute phase in the ICU. | The early acute phase is between 24 and 72 hours after ICU admission, and the late acute phase between 120 and 148 hours, i.e., 5-7 days after ICU admission.
  Difference in endogenous rate of appearance, calculated from enrichment of labelled substrates in plasma glycerol, between the fasted and fed state in the early acute phase, compared to the late acute phase in the ICU.
Attenuation of phenylalanine production in response to nutrition in the late acute phase compared to the early acute phase in the ICU. | The early acute phase is between 24 and 72 hours after ICU admission, and the late acute phase between 120 and 148 hours, i.e., 5-7 days after ICU admission.
  Difference in endogenous rate of appearance, calculated from enrichment of labelled substrates in plasma phenylalanine, between the fasted and fed state in the early acute phase, compared to the late acute phase in the ICU.
Attenuation of glucose production in response to nutrition in the early acute phase in the ICU compared to healthy controls. | Early acute phase of critical illness, i.e., 24-72 hours after ICU admission. The difference between substrate kinetics at 165-180 min and 345-360 min after the start of the tracer infusion will be calculated.
  Difference in endogenous rate of appearance, calculated from enrichment of labeled substrates in plasma of glucose between fasted and fed state in the early acute phase, compared to healthy controls.
Attenuation of glycerol production in response to nutrition in the early acute phase in the ICU compared to healthy controls. | Early acute phase of critical illness, i.e., 24-72 hours after ICU admission. The difference between substrate kinetics at 165-180 min and 345-360 min after the start of the tracer infusion will be calculated.
  Difference in endogenous rate of appearance, calculated from enrichment of labelled substrates in plasma of glycerol between fasted and fed state in the early acute phase, compared to healthy controls.
Attenuation of phenylalanine production in response to nutrition in the early acute phase in the ICU compared to healthy controls. | Early acute phase of critical illness, i.e., 24-72 hours after ICU admission. The difference between substrate kinetics at 165-180 min and 345-360 min after the start of the tracer infusion will be calculated.
  Difference in endogenous rate of appearance, calculated from enrichment of labelled substrates in plasma of phenylalanine between fasted and fed state in the early acute phase, compared to healthy controls.
Difference in non-suppressible glucose production in the fed state between ICU patients. | The early acute phase is between 24 and 72 hours after ICU admission, and the late acute phase between 120 and 148 hours, i.e., 5-7 days after ICU admission.
  Mean change in endogenous rate of appearance, calculated from enrichment of labelled substrates in plasma of glucose between the fasted and fed state in the early acute phase compared to the late acute phase.
Difference in non-suppressible glycerol production in the fed state between ICU patients. | The early acute phase is between 24 and 72 hours after ICU admission, and the late acute phase between 120 and 148 hours, i.e., 5-7 days after ICU admission.
  Mean change in endogenous rate of appearance, calculated from enrichment of labelled substrates in plasma of glycerol between the fasted and fed state in the early acute phase compared to the late acute phase.
Difference in non-suppressible phenylalanine production in the fed state between ICU patients. | The early acute phase is between 24 and 72 hours after ICU admission, and the late acute phase between 120 and 148 hours, i.e., 5-7 days after ICU admission.
  Mean change in endogenous rate of appearance, calculated from enrichment of labelled substrates in plasma of phenylalanine between the fasted and fed state in the early acute phase compared to the late acute phase.

OTHER OUTCOMES:
Metabolomics | The early acute phase is between 24 and 72 hours after ICU admission, and the late acute phase is between 120 and 148 hours, i.e., 5-7 days after ICU admission.
  Within-group changes in ICU patients between the fasted and fed states of metabolomics. This will be compared between the early acute and the late acute phase.
Attenuation of glucose production in response to nutrition in the late phase compared to the early acute phase in the ICU. | The early acute phase is between 24 and 72 hours after ICU admission, and the late acute phase is more than 240 hours, i.e., 10 days after ICU admission.
  Difference in endogenous rate of appearance, calculated from enrichment of labelled substrates in plasma of glucose between fasted and fed states in the early acute phase, compared to the late phase in the ICU.
Attenuation of glycerol production in response to nutrition in the late phase compared to the early acute phase in the ICU. | The early acute phase is between 24 and 72 hours after ICU admission, and the late acute phase is more than 240 hours, i.e., 10 days after ICU admission.
  Difference in endogenous rate of appearance, calculated from enrichment of labelled substrates in plasma of glycerol between fasted and fed states in the early acute phase, compared to the late phase in the ICU.
Attenuation of phenylalanine production in response to nutrition in the late phase compared to the early acute phase in the ICU. | The early acute phase is between 24 and 72 hours after ICU admission, and the late acute phase is more than 240 hours, i.e., 10 days after ICU admission.
  Difference in endogenous rate of appearance, calculated from enrichment of labelled substrates in plasma of phanylalanine between fasted and fed states in the early acute phase, compared to the late phase in the ICU.
Changes in insulin levels | The early acute phase is between 24 and 72 hours after ICU admission, and the late acute phase is between 120 and 148 hours, i.e., 5-7 days after ICU admission.
  Within-group changes in ICU patients between the fasted and fed states of insulin. This will be compared between the early acute and the late acute phase.
Changes in C-peptide levels | The early acute phase is between 24 and 72 hours after ICU admission, and the late acute phase is between 120 and 148 hours, i.e., 5-7 days after ICU admission.
  Within-group changes in ICU patients between the fasted and fed states of C-peptide. This will be compared between the early acute and the late acute phase.
Changes in glucagon levels | The early acute phase is between 24 and 72 hours after ICU admission, and the late acute phase is between 120 and 148 hours, i.e., 5-7 days after ICU admission.
  Within-group changes in ICU patients between the fasted and fed states of glucagon. This will be compared between the early acute and the late acute phase.
Changes in C-reactive protein levels. | The early acute phase is between 24 and 72 hours after ICU admission, and the late acute phase is between 120 and 148 hours, i.e., 5-7 days after ICU admission.
  Within-group changes in ICU patients between the fasted and fed states of C-reactive protein. This will be compared between the early acute and the late acute phase.
Changes in cytokine levels. | The early acute phase is between 24 and 72 hours after ICU admission, and the late acute phase is between 120 and 148 hours, i.e., 5-7 days after ICU admission.
  Within-group changes in ICU patients between the fasted and fed states of cytokines. This will be compared between the early acute and the late acute phase.
Changes in urea levels. | The early acute phase is between 24 and 72 hours after ICU admission, and the late acute phase is between 120 and 148 hours, i.e., 5-7 days after ICU admission.
  Within-group changes in ICU patients between the fasted and fed states of urea. This will be compared between the early acute and the late acute phase.
Changes in free amino acids levels. | The early acute phase is between 24 and 72 hours after ICU admission, and the late acute phase is between 120 and 148 hours, i.e., 5-7 days after ICU admission.
  Within-group changes in ICU patients between the fasted and fed states of free amino acids. This will be compared between the early acute and the late acute phase.
Changes in triglyceride levels. | The early acute phase is between 24 and 72 hours after ICU admission, and the late acute phase is between 120 and 148 hours, i.e., 5-7 days after ICU admission.
  Within-group changes in ICU patients between the fasted and fed states of triglycerides. This will be compared between the early acute and the late acute phase.
Changes in free fatty acid levels. | The early acute phase is between 24 and 72 hours after ICU admission, and the late acute phase is between 120 and 148 hours, i.e., 5-7 days after ICU admission.
  Within-group changes in ICU patients between the fasted and fed states of free fatty acids. This will be compared between the early acute and the late acute phase.

CONTACTS AND LOCATIONS:
Overall Officials: Olav Rooyackers, PhD, Study Chair — Karolinska University Hospital/Karolinska Institute; Martin Sundström Rehal, MD PhD, Principal Investigator — Karolinska University Hospital/Karolinska Institute
Locations (1):
- Karolinska University Hospital Huddinge, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
IPD will not be routinely shared due to patient confidentiality. Anonymized parts of the data set may be shared on reasonable request.